CLINICAL TRIAL: NCT07209969
Title: Efficacy of Cognitive Behaviour Therapy for Insomnia (CBT-I) in Adolescents With Attention Deficit Hyperactivity Disorder (ADHD): a Randomised Controlled Trial
Brief Title: CBT-I in Adolescents With ADHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Kwai Chung Hospital (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KW/FR-21-131(163-09)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Insomnia; ADHD
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-I group (Experimental): The intervention for the CBT-I group will involve five weekly 60-minute individual, face-to-face sessions of CBT-I. The treatment components aim to address the behavioural, cognitive and physiological perpetuating factor of insomnia whilst considering the clinical context of ADHD and include: psychoeducation about sleep, circadian rhythm, sleep hygiene, sleep restriction, stimulus control, cognitive restructuring, and relaxation techniques.
  Interventions: Behavioral: CBT-I group
- TAU group (No Intervention): Participants will continue their usual clinical follow-up and receive standard treatment at the clinic.

INTERVENTIONS:
Behavioral: CBT-I group — Refer to the arm description
  Arms: CBT-I group

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is a neurodevelopmental disorder characterized by persistent patterns of inattention, hyperactivity, and impulsivity, affecting individuals across the lifespan. While the core symptoms of ADHD are well-documented, emerging research has shed light on the prevalence of comorbid sleep disturbances, particularly insomnia, among adolescents with ADHD. The co-occurrence of ADHD and insomnia can exacerbate cognitive and emotional difficulties, impacting various aspects of daily functioning. Cognitive-Behavioral Therapy for Insomnia (CBT-I) has proven effective in addressing sleep-related difficulties in various populations. However, there is a paucity of research specifically examining the efficacy of CBT-I in adolescents with ADHD. To date, there was only one pilot single-arm sleep intervention study conducted in adolescents with ADHD (Becker et al., 2021) and one randomized controlled trial of sleep intervention in adolescents with ADHD that is still undergoing data collection (Keuppens et al., 2023). Given the lack of research on the intervention for insomnia in the context of ADHD, this study aimed to evaluate the efficacy of CBT-I on adolescents with ADHD in insomnia symptoms, sleep related cognitions and practices, ADHD severity, emotion regulation ability, and depressive and anxiety symptoms.

DETAILED DESCRIPTION:
An assessor-blind, parallel-group, randomised controlled trial will be conducted in adolescents with comorbid ADHD and insomnia. Eligible participants will be randomised to either CBT-I group (intervention) or treatment-as-usual (TAU) control group. Assessments will be conducted at baseline, one-week post-treatment, and post-treatment 3-month. During the study period, all the participants will continue their regular clinical follow-ups with their attending psychiatrist for the prescription of psychotropic medication(s), if needed, for managing their ADHD and mental health condition. Prescription of any psychotropic medications of each participant during the trial will be reviewed and documented at baseline and at each follow-up.

ELIGIBILITY:
Inclusion Criteria: Adolescents aged 11-18 years old meeting the following inclusion criteria were invited to take part in the present study:

1. Having a clinical diagnosis of ADHD made by health care professionals (psychiatrist, clinical psychologist, or educational psychologist) based on self-report;
2. a DSM-5 diagnosis of insomnia disorder, and a score on ISI ≥ 9 (suggested cut-off for adolescents) (Chung et al., 2011);
3. Those who agreed to keep the same dosage of medication throughout the study up till completion of follow up assessments.

Exclusion Criteria: Adolescents were excluded if they met any of the following criteria:

1. A current diagnosis of substance abuse or dependence; a current or past history of manic or hypomanic episode, schizophrenia spectrum disorders, autism spectrum disorders, organic mental disorders, or intellectual disabilities;
2. Having a prominent medical condition known to interfere with sleep continuity and quality (e.g. severe eczema, gastro-oesophageal reflux disease);
3. Having a clinically diagnosed sleep disorder that may potentially contribute to a disruption in sleep continuity and quality, such as narcolepsy, sleep-disordered breathing, and restless leg syndrome, based on self-reported medical history;
4. On an optimal dosage of psychostimulant or nonstimulant ADHD medications for less than a month;
5. Concurrent, regular use of psychotropic medications(s) known to affect sleep continuity and quality (e.g. hypnotics, steroids), except for the use of psychostimulant medication for ADHD;
6. Receiving ongoing pharmacological and psychological treatment for insomnia;
7. With hearing or speech deficit.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in insomnia symptoms | Baseline, one-week post-treatment and 3 month post-treatment
  Insomnia symptoms measured by Insomnia Severity Index (ISI). ISI is a 5-item self-rated scale. Possible scores range from 0 to 20, with higher scores indicating higher insomnia severity.

SECONDARY OUTCOMES:
Change in individual beliefs and attitude about sleep | Baseline, one-week post-treatment and 3 month post-treatment
  Dysfunctional Beliefs and Attitudes about Sleep (DBAS) is a 16-item self-rated scale measuring the respondent's sleep-related beliefs, more specifically, their expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues. A total score is calculated by averaging score of all items, possibly scored 0 to 10, with a higher score indicating more dysfunctional beliefs and attitudes about sleep.
Change in adolescent sleep hygiene | Baseline, one-week post-treatment and 3 month post-treatment
  The Revised Adolescents Sleep Hygiene Scale (ASHSr) is used to measure adolescent sleep hygiene. It comprises 33 self-report items, categorizing into six subscales: physiological, sleep environment, cognitive/emotional, sleep stability, daytime sleep, and behavioral arousal. Adolescents rate the frequency of their sleep-related behaviors over the past month using a 6-point scale, where 1 corresponds to "always" and 6 to "never." Subscale scores are computed using means, and these scores range from 1 to 6. Higher scores on the subscales indicate better sleep hygiene.
Change in ADHD symptoms (Self-report) | Baseline, one-week post-treatment and 3 month post-treatment
  The Adult ADHD Self-Report Scale (ASRS) v1.1 Symptom Checklist is an 18-item self-administered questionnaire to screen for ADHD symptoms in both community surveys and clinical settings based on criteria of the DSM-IV-TR. The questionnaire asks participants to rate how often a symptom of inattention or hyperactivity has occurred during the past 6 months using a scale from 0 (never) to 4 (very often). The total score on this scale can range from 0 to 72, with higher scores indicating more ADHD symptomology.
Change in anxiety symptoms | Baseline, one-week post-treatment and 3 month post-treatment
  The Generalized Anxiety Disorder 7-item scale (GAD-7) will be used to measure generalized anxiety symptoms in the past 2 weeks
Change in depressive symptoms | Baseline, one-week post-treatment and 3 month post-treatment
  The Patient Health Questionnaire - 9 (PHQ-9) will be used to measure the presence and severity of depression in the past 2 weeks.
Change in emotion regulation ability | Baseline, one-week post-treatment and 3 month post-treatment
  The Difficulty in Emotion Regulation Scale (DERS; (Gratz & Roemer, 2004) will be used to assess six domains of emotion regulation ability.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Child and adolescent outpatient psychiatric clinic of Kwai Chung Hospital, Hong Kong
  - Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No